CLINICAL TRIAL: NCT02129686
Title: A Randomized Pilot Study of Acupuncture for Chemotherapy-induced Peripheral Neuropathy in Breast Cancer Patients
Brief Title: A Pilot Study of Acupuncture for Chemotherapy-induced Peripheral Neuropathy in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: The Comprehensive and Integrative Medicine Institute of South Korea (Other)
Responsible Party: Principal Investigator, Weidong Lu, MB, MPH, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-067
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Taxane-induced Peripheral Neuropathy; Chemotherapy-induced Peripheral Neuropathy (CIPN); Early-Stage Breast Carcinoma; Stage I Breast Cancer; Stage II Breast Cancer; Stage III Breast Cancer
Keywords: Chemotherapy-induced peripheral neuropathy (CIPN); Acupuncture; Early-Stage Breast Carcinoma; Stage I Breast Cancer; Stage II Breast Cancer; Stage III Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Acupuncture Group (Experimental): Immediate acupuncture arm will receive acupuncture 3 times per week during week 1 and week 2, then 2 times per week from week 2 to week 8 for a total of 18 sessions. The crossover will take place after 8th week.
  The immediate acupuncture arm will enter a follow-up phase without acupuncture for 8 weeks from week 9 to week 16, while the standard usual care will be provided.
  Interventions: Procedure: Immediate Acupuncture Group
- Delayed Acupuncture Group (Active Comparator): The patients on the usual care/delayed acupuncture arm will continue their standard usual care with their physicians and care team. The crossover will take place after 8th week. After crossover, the patients initially on the usual care/delayed acupuncture arm will receive the identical acupuncture protocol but a less frequent schedule from week 9 to week 16: 2 times per week at week 9, then 1 time per week from week 10 to week 16 for a total of 9 sessions
  Interventions: Procedure: Delayed Acupuncture Group

INTERVENTIONS:
Procedure: Immediate Acupuncture Group
  Arms: Immediate Acupuncture Group
Procedure: Delayed Acupuncture Group
  Arms: Delayed Acupuncture Group

SUMMARY:
This study is being done to evaluate the potential benefits of using acupuncture to reduce symptoms of tingling, burning, numbness and pain in the hands and feet of women with peripheral neuropathy after completion of chemotherapy for breast cancer.

DETAILED DESCRIPTION:
Chemotherapy drugs used to treat cancer can cause temporary or permanent damage to the nerves in the hands and feet, a condition called "chemotherapy-induced peripheral neuropathy". The most common symptoms of chemotherapy-induced peripheral neuropathy are pain, tingling, burning or numbness sensation, which can lead to balance problems or trouble using fingers or pick up/holding things. These symptoms often last months to years after the completion of chemotherapy. Medications and nutritional supplements can ease the symptoms of chemotherapy-induced peripheral neuropathy, but many patients continue to experience symptoms despite these treatments.

Acupuncture is an intervention in which hair-thin, stainless steel needles are shallowly inserted into specific points on the skin, with the goal of influencing the body's natural healing system. Acupuncture has been studied in clinical trials in cancer patients and has been shown to be effective for various conditions including chemotherapy-induced nausea and vomiting. A few preliminary studies have suggested that acupuncture may help to reduce symptoms of peripheral neuropathy, but more information is needed about the benefits of acupuncture in breast cancer patients This study is being done to evaluate the potential benefits of using acupuncture to reduce symptoms of tingling, burning, numbness and pain in the hands and feet of women with peripheral neuropathy after completion of chemotherapy for breast cancer.

This research study will help to determine the benefits of acupuncture for the treatment of chemotherapy-induced peripheral neuropathy. The study will also look at two different acupuncture schedules to determine whether patients derive benefits from lower and higher dose acupuncture treatments.

ELIGIBILITY:
Inclusion Criteria:

* History of histologically or cytologically proven breast cancer at stage I, II and III, without evidence of distant metastasis;
* Completed adjuvant taxane-based chemotherapy as single agents or in combination with platins or HER-2 directed therapy
* Reporting grade 1 or greater of the following symptoms persistently for more than 2 weeks: neuropathic pain, allodynia, areflexia, dysesthesia, paresthesia, hyperesthesia, hypoesthesia or glove and stocking syndrome as defined by Common Terminology Criteria for Adverse Events (CTCAE v. 4.03) (Table 1 and the screening checklist);
* Patients who are currently on stable prescription medications or dietary supplements for CIPN and still symptomatic as defined above will be allowed to participate in the study. Related medications are: gabapentin, pregabalin, nortriptyline, amitriptyline, duloxetine, venlafaxine; lidocaine, opioid tramadol and other narcotics; NSAIDs; glutamine, glutathione, vitamin E and vitamin B12;
* Age ≥ 18 years;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Adequate hematological function: neutrophil count >1.0 x109/L, platelet count >50x109/L;
* Signed informed consent.

Exclusion Criteria:

* Patients with any of the following criteria will not be eligible for the study:
* Unstable cardiac disease or myocardial infarction within 6 months prior to study entry;
* Wearing a pacemaker or implantable cardioverter-defibrillator; uncontrolled seizure disorder;
* History of pre-existing peripheral neuropathy prior to chemotherapy, including alcoholism, vitamin B deficiency, diabetes, HIV, congenital neuropathy, toxic neuropathy;
* Peripheral neuropathy caused by tumor infiltration or compression of spinal nerves or surgical trauma;
* Pregnancy or potential pregnancy and nursing;
* Active clinically significant uncontrolled infection;
* Prior use of acupuncture for CIPN within 6 months prior to study entry;
* Patients with uncontrolled major psychiatric disorders, such as major depression or psychosis, will not be eligible for this trial. Patients with a history of depression or anxiety who are stable on or off psychiatric medications will be eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Response Rate from Baseline in PNQ Score | Baseline, Week 8
  The PNQ includes two questionnaire items: one asking about sensory neurotoxicity and the other asking about motor neurotoxicity. The questionnaire items correspond to the neurotoxicity questions included in the NCI-CTCAE. PNQ grades range from grade A (no neuropathy) to grade E (very severe neuropathy). Answer options will be coded 0=A to 4=E, with a higher score indicating more severe CIPN

SECONDARY OUTCOMES:
Changes in FACT/NTX subscale baseline to 8 weeks | Baseline, 8 Weeks
Changes in EORTC-QLQ-CIPN20 subscale Baseline, 8 Weeks | Baseline, 8 Weeks
  Comprised of three subscales assessing sensory, motor, and autonomic symptoms. Subscale scores will be calculated and linearly transformed to a 0 to 100 scale, with higher scores suggesting more severe symptoms. Changes from baseline (8-week - baseline) between the intervention arms for each subscale will be of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Lu, M.B., MPH, Ph.D, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lu W, Giobbie-Hurder A, Freedman RA, Shin IH, Lin NU, Partridge AH, Rosenthal DS, Ligibel JA. Acupuncture for Chemotherapy-Induced Peripheral Neuropathy in Breast Cancer Survivors: A Randomized Controlled Pilot Trial. Oncologist. 2020 Apr;25(4):310-318. doi: 10.1634/theoncologist.2019-0489. Epub 2019 Oct 14. PMID 32297442
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7160396/